CLINICAL TRIAL: NCT05141175
Title: The Duke Primary Care Tailored to You (TTY) Blood Pressure Control Pilot Study
Brief Title: Tailored to You (TTY) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00109188
Record Dates: First submitted 2021-11-15; First posted 2021-12-02 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Cardiography, Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypertension patients (Experimental): Patients with documented diagnosis of hypertension and their most recent office systolic BP average measured using automated office BP is ≥140 mmHg systolic or ≥90 mmHg diastolic and they are currently prescribed at least one BP-lowering medication will be recruited.
  Interventions: Device: Hypertension medication algorithm; Device: Impedance Cardiography

INTERVENTIONS:
Device: Hypertension medication algorithm — The algorithm is configured to align medication choices based on the hemodynamic findings from the ICG readings. This decision support tool was created so as to organize these medications based on their mechanism of action and is consistent with the evidence-based treatment of hypertension.
Device: Impedance Cardiography — The ICG system provides a printed report that indicates whether a person's hemodynamic state is predominantly one that is vasoconstricted, hyperdynamic, or mixed

SUMMARY:
The purpose of this research study is to use a test called impedance cardiography (ICG) to provide more information about how to improve the control of blood pressure. Participants will be given this test so investigators can get more information about what is going on inside the heart and blood vessels that is contributing to high blood pressure. ICG is a lot like an EKG (electrocardiogram) in that it uses electrodes and a computer to make a report. Participants will lie down on the exam table and two electrodes go on the right ankle and two electrodes go on the left wrist. The process takes about 5 minutes and is painless and not invasive.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of hypertension
* Most recent office systolic BP average measured using automated office BP (AOBP) is ≥140 mmHg systolic or ≥90 mmHg diastolic
* Currently prescribed at least one BP-lowering medication
* Under the care of a primary care clinician

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Viera, MD, Principal Investigator — Duke University
Locations (1):
- Duke Primary Care, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypertension Patients
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled as Measured by Enrollment Logs
Time Frame: 1.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Number of Participants That Completed Study as Measured by Enrollment Logs
Time Frame: 1.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 20
Participants | 19

3. Secondary Outcome: Change in Blood Pressure as Measured by Medical Record
Time Frame: Baseline, 4 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 19
mmHg
  systolic blood pressure | 11 (7)
  diastolic blood pressure | 3 (3)

4. Secondary Outcome: Number of Anti-hypertensive Medications Prescribed as Measured by Medical Record Review
Time Frame: Up to 4 months
Measure: Mean (Standard Deviation); unit: anti-hypertensive medications
Arm/Group | Hypertension Patients
Number analyzed (Participants) | 19
anti-hypertensive medications | 2.60 (.5)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Hypertension Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT05141175/Prot_001.pdf